CLINICAL TRIAL: NCT01179776
Title: A Single Center, Open, Randomized, Placebo-controlled Study Investigating the Safety of Administration of Ilomedin® in Addition to Standard Treatment in Patients Having Undergone Primary Percutaneous Coronary Intervention (PCI)
Brief Title: Ilomedin Treatment for Patients Having Undergone Primary Percutaneous Coronary Intervention (PCI)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Thrombologic ApS (Industry)
Collaborators: Lene Holmvang (Unknown); Rigshospitalet, Denmark (Other)
Responsible Party: Lene Holmvang, Rigshospitalet
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: THR-PS-02
Record Dates: First submitted 2010-08-10; First posted 2010-08-11 (Estimated); Last update posted 2011-06-02 (Estimated); Status verified 2011-06

CONDITIONS: Myocardial Infarct
Keywords: ST-eleveation; Myocardial infarct; Percutaneous coronary intervention; Myocardial infarct STEMI patients
MeSH Terms: conditions — Myocardial Infarction | interventions — Iloprost; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ilomedin and standard low dose treatment (Experimental)
  Interventions: Drug: Ilomedin; Drug: Ilomedin and standard low dose treatment
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ilomedin — Ilomedin
  Other Names: Iloprost
  Arms: Ilomedin and standard low dose treatment
Drug: Placebo — i.v saline
  Arms: Placebo
Drug: Ilomedin
  Arms: Ilomedin and standard low dose treatment
Drug: Ilomedin and standard low dose treatment
  Arms: Ilomedin and standard low dose treatment

SUMMARY:
Acute myocardial infarct patients with STEMI (ST-elevation on ECG) whom undergo a primary percutaneous cardiac intervention will following the standard treatment , received low dose of Ilomedin and to low dose of standard treatment for another 24 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Undergoing primary PCI due to STEMI (TIMI flow I -III before PCI and symptom duration < 12 hours)

6) Following receipt of verbal and written information about the study, the patient must provide signed informed consent before any study data is used.

-

Exclusion Criteria:

2) Not able to give informed consent 3) Women with childbearing potential 4) On-going concomitant treatment with K-vitamin antagonists (one bolus dose pre-PCI allowed) 5) Known congenital or acquired coagulopathy and/or thrombocytopathy s 8) Participation in a clinical study and/or another investigational device within the past four weeks prior to Day 1 9) Major surgery or trauma within the past 6 weeks prior to Day 1 10) A blood coagulation disorder (i.e. international normalized ratio [INR] > 2.0, platelet count < 100,000/mm3, or hematocrit < 30%) 11) Renal insufficiency (creatinine > 140 mmol/l) 12) Major procedure related bleeding (TIMI major criteria); GI or urinary tract bleeding prior to inclusion in the trial 13) Known active hepatitis B and/or hepatitis C or HIV 14) Known or suspected hypersensitivity to components of the investigational medicinal product

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-09; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Bleeding complications as evaluated by TIMI and GUSTO criteria | Feb 2011
  Increased bleeding complications will be evaluated between the active and placebo groups.

SECONDARY OUTCOMES:
Endothelial markers and blood aggregation (measured by TEG and multiplate) | Feb 2011
  Endothelial markers will be measured to evaluate the Ilomedin effect on these patients. Blood aggregation and coagulation will be evaluated by using TEG and Multiplate.

CONTACTS AND LOCATIONS:
Overall Officials: Lene Holmvang, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Lene Holmvang, Copenhagen, Denmark

REFERENCES:
- [Derived] Holmvang L, Ostrowski SR, Dridi NP, Johansson P. A single center, open, randomized study investigating the clinical safety and the endothelial modulating effects of a prostacyclin analog in combination with eptifibatide in patients having undergone primary percutaneous coronary intervention (PCI) for ST-segment elevation myocardial infarction. Prostaglandins Other Lipid Mediat. 2012 Dec;99(3-4):87-95. doi: 10.1016/j.prostaglandins.2012.08.002. Epub 2012 Aug 28. PMID 22951358